CLINICAL TRIAL: NCT01704365
Title: A Phase II Randomized, Observer-Blinded, Placebo-Controlled, Dose-Ranging Study to Evaluate the Immunogenicity and Safety of an RSV-F Protein Nanoparticle Vaccine, With or Without Aluminum, in Healthy Women of Child-Bearing Age
Brief Title: RSV-F Vaccine Dose Ranging Study in Young Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novavax (Industry)
Collaborators: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NVX757.201
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-02

CONDITIONS: Respiratory Syncytial Virus (RSV)
MeSH Terms: interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- Group A (Experimental): Low dose RSV-F Vaccine with Adjuvant (Day 0 and Day 28)
  Interventions: Biological: Low dose RSV-F Vaccine with Adjuvant
- Group B (Experimental): Low dose RSV-F Vaccine with Adjuvant (Day 0); Placebo (Day 28)
  Interventions: Biological: Low dose RSV-F Vaccine with Adjuvant; Biological: Placebo
- Group C (Experimental): Low dose RSV-F Vaccine without Adjuvant (Day 0 and Day 28)
  Interventions: Biological: Low dose RSV-F Vaccine without Adjuvant
- Group D (Experimental): Low dose RSV-F Vaccine without Adjuvant (Day 0); Placebo (Day 28)
  Interventions: Biological: Low dose RSV-F Vaccine without Adjuvant; Biological: Placebo
- Group E (Experimental): High dose RSV-F Vaccine with Adjuvant (Day 0 and Day 28)
  Interventions: Biological: High dose RSV-F Vaccine with Adjuvant
- Group F (Experimental): High dose RSV-F Vaccine with Adjuvant (Day 0); Placebo (Day 28)
  Interventions: Biological: High dose RSV-F Vaccine with Adjuvant; Biological: Placebo
- Group G (Experimental): High dose RSV-F Vaccine without Adjuvant (Day 0 and Day 28)
  Interventions: Biological: High dose RSV-F Vaccine without Adjuvant
- Group H (Experimental): High dose RSV-F Vaccine without Adjuvant (Day 0); Placebo (Day 28)
  Interventions: Biological: High dose RSV-F Vaccine without Adjuvant; Biological: Placebo
- Group J (Experimental): Low dose RSV-F Vaccine with Adjuvant [Bedside Mixing] (Day 0 & Day 28)
  Interventions: Biological: Low dose RSV-F Vaccine with Adjuvant [Bedside Mixing]
- Group K (Placebo Comparator): Placebo (Day 0 and Day 28)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Low dose RSV-F Vaccine with Adjuvant — 0.5mL IM Injection
  Arms: Group A; Group B
Biological: Low dose RSV-F Vaccine without Adjuvant — 0.5ml IM Injection
  Arms: Group C; Group D
Biological: High dose RSV-F Vaccine with Adjuvant — 0.5mL IM Injection
  Arms: Group E; Group F
Biological: High dose RSV-F Vaccine without Adjuvant — 0.5mL IM Injection
  Arms: Group G; Group H
Biological: Low dose RSV-F Vaccine with Adjuvant [Bedside Mixing] — 0.5mL IM Injection
  Arms: Group J
Biological: Placebo — 0.5mL IM Injection
  Arms: Group B; Group D; Group F; Group H; Group K

SUMMARY:
The purpose of this study is to evaluate the immunogenicty and safety of an RSV-F protein nanoparticle vaccine, with out without aluminum, in healthy women of child-bearing potential.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult females, ≥ 18 and ≤ 35 years of age. "Healthy" shall be defined by the absence of any illness, acute or chronic, that requires ongoing systemic therapy for the control of symptoms or prevention of disability.
* Subjects on stable (no change in ≥ 3 months) therapy for findings (e.g., hypertension or hyperlipidemia) that are not associated with symptoms or disability are eligible, as are users of hormonal contraceptives.
* Subjects who receive intermittent prophylaxis for risks associated with asymptomatic findings (e.g., antibiotic prophylaxis prior to dental procedures in a subject with mitral valve prolapse) are eligible.
* Ongoing therapy will be defined as continuous or, if intermittent, more frequent than once every 3 months (e.g., use of an inhaled bronchodilator for exercise-induced bronchospasm more than once every 3 months). Immunosuppressives are subject to exclusion criterion #5 below.
* Persons being treated for illnesses or conditions that would become acutely symptomatic or disabling in the absence of treatment are not eligible.
* Willing and able to give informed consent prior to study enrollment.
* Able to comply with study requirements.
* Women who are not surgically sterile must have a negative urine pregnancy test prior to each vaccination; will be advised through the Informed Consent process to avoid becoming pregnant over the duration of the study, and must assert that they will employ an effective form of birth control for the duration of the study. Acceptable forms of birth control are: credible history of continuous abstinence from heterosexual activity, hormonal contraceptives (oral, injectable, implant, patch, ring), double-barrier contraceptives (condom or diaphragm, with spermicide), and IUD.

Exclusion Criteria:

* Participation in research involving investigational product (drug / biologic / device) within 45 days before planned date of first vaccination.
* History of a serious reaction to any prior vaccination.
* Received any vaccine in the 4 weeks preceding the study vaccination; or any RSV vaccine at any time.
* Any known or suspected immunosuppressive condition, acquired or congenital, as determined by history and/or physical examination.
* Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the study vaccine. An immunosuppressant dose of glucocorticoid will be defined as a systemic dose ≥10mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids will be permitted.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study vaccine or during the study.
* Acute disease at the time of enrollment (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature >38.0°C on the planned day of vaccine administration).
* Known disturbance of coagulation.
* Women who are pregnant or breastfeeding, or plan to become pregnant during the study.
* Suspicion or recent history (within one year of planned vaccination) of alcohol or other substance abuse.
* Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled or could interfere with evaluation of the vaccine or interpretation of study results (including neurologic or psychiatric conditions deemed likely to impair the quality of safety reporting).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 330 (Actual)
Dates: Start 2012-10; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Immunogenicity as assessed by serum IgG antibody titers specific for the F-Protein antigen across treatment groups | Day 0 to Day 112
  Immunogenicity will be measured using derived / calculated endpoints based on:
  * Geometric mean titer (GMT)
  * Geometric mean ratio (GMR)
  * Seroconversion rate (SCR)
  * Seroresponse rate (SRR)
Assessment of the safety | Day 0 to Day 182
  Number (and percentage) of subjects with solicited local and systemic Adverse Events over the seven days post-injections; all adverse events, solicited and unsolicited over 56 days post-first injection.
  Significant New Medical Conditions, Medically Attended Events and Serious Adverse Events will be collected for six months

SECONDARY OUTCOMES:
Immunogenicity based on neturalizing antibody titer | Day 0 to Day 112

CONTACTS AND LOCATIONS:
Overall Officials: D. Nigel Thomas, Ph.D., Study Director — Novavax, Inc.
Locations (4):
- United States (4):
  - Anaheim Clinical Trials, Anaheim, California
  - Accelovance Rockville, Rockville, Maryland
  - Coastal Carolina Research, Mt. Pleasant, South Carolina
  - Clinical Trials of Texas, San Antonio, Texas

REFERENCES:
- [Derived] Glenn GM, Fries LF, Thomas DN, Smith G, Kpamegan E, Lu H, Flyer D, Jani D, Hickman SP, Piedra PA. A Randomized, Blinded, Controlled, Dose-Ranging Study of a Respiratory Syncytial Virus Recombinant Fusion (F) Nanoparticle Vaccine in Healthy Women of Childbearing Age. J Infect Dis. 2016 Feb 1;213(3):411-22. doi: 10.1093/infdis/jiv406. Epub 2015 Aug 10. PMID 26259809
- See also: Novavax Homepage — http://www.novavax.com